CLINICAL TRIAL: NCT02484716
Title: Efficacy of a Timolol Nasal Spray as a Treatment for Epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT) - Randomized Trial Versus Placebo
Brief Title: Efficacy of a Timolol Nasal Spray as a Treatment for Epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT) - (TEMPO)
Acronym: TEMPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL15_0063; 2015-000385-55 (EudraCT Number)
Record Dates: First submitted 2015-06-17; First posted 2015-06-30 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic; Osler Rendu Disease
Keywords: Hereditary Hemorrhagic Telangiectasia (HHT); Antiangiogenic therapy; Timolol
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Timolol (Experimental): Timolol 0.5% eye-drops solution packaged in a nasal spray device.
  Interventions: Drug: Timolol nasal spray
- Placebo (Placebo Comparator): NaCl solution packaged in a nasal spray device.
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Timolol nasal spray — Timolol 0.5% is administered by the patient with a posology of one spray (50 µL) in each nostril twice a day for 4 weeks.
  Arms: Timolol
Drug: Placebo nasal spray — Placebo (NaCl) is administered by the patient with a posology of one spray (50 µL) in each nostril twice a day for 4 weeks.
  Arms: Placebo

SUMMARY:
Timolol is a nonselective β-blocker commonly used in the treatment of glaucoma. Recently it has been used topically for the treatment of superficial hemangiomas. Because of its potential mechanism of action, it is possible that timolol could also be useful for the treatment of epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT). Moreover a case was reported in 2012 showing an improvement of nosebleeds with the use of topical nasal timolol. The aim of the study is to evaluate timolol nasal spray efficacy in HHT.

The main objective of this trial is to evaluate, 3 months after the end of the treatment, the efficacy on the duration of nosebleeds of a 4 weeks timolol intranasal treatment in HHT patients with nosebleeds (>20 min/month). Secondary objectives are to evaluate the tolerance, the efficacy at 6 months after the end of the treatment, and the efficacy on anemia and on clinical parameters (nosebleeds, quality of life and blood transfusions).

This is a prospective double blind phase II study, randomized versus placebo using an allocation ratio of 1:1. A total of 58 patients will be included. The product (solution with timolol at 0.5% or placebo) is self-administered by the patient with a posology of one spray (50 µL) in each nostril twice a day for 28 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients who give voluntary, informed consent and sign a consent form.
* Patients affiliated with the French universal health care system
* Patients treated for HHT, that has been confirmed clinically (presence of at least 3 Curaçao criteria) and/or by molecular biology.
* Patients who present epistaxis averaging over 20 minutes in the three months before inclusion, justified by completed epistaxis tally sheets.

Exclusion Criteria:

* Pregnant women or women who could become pregnant during the study, or during lactation
* Patients not affiliated with the French universal health care system
* Patients who are protected adults according to the terms of the law (French public health laws).
* Refusal to give consent.
* Patients whose HHT diagnosis has not be confirmed clinically and/or by molecular biology.
* Participation in another therapeutic trial which could interfere with the present trial (investigator jugement).
* Bronchial asthma, presence or history of severe chronic obstructive pulmonary disease
* Cardiac history : cardiac failure or cardiogenic shock. Atrioventricular block (second or third degrees) not controlled with pace-maker or sinus disease (included sinoatrial block) confirmed by ECG less than one year. Ongoing treatment by calcium antagonists (bépridil, diltiazem, verapamil) or antiarrhytmics (propafénone, quinidine, hydroquinidine, disopyramide) or clonidine or lidocaîne. Ongoing beta-blocker treatment.
* Bradycardia (<50 pulse per minute)
* Hypotension (PAS < 90 Hg mm)
* Angina
* Not controlled Pheochromocytoma
* Severe peripheral circulatory disturbances (Raynaud disease)
* Hypersensitivity to the active substance, any of the excipients or other beta-blocking agents
* Ongoing treatment by floctafénine or sultopride or amiodarone
* Patients who do not complete epistaxis grids for three months before treatment
* Patients who present epistaxis averaging below 20 minutes in the three months before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Efficacy of timolol nasal spray on duration of nosebleeds for 3 months after the end of the treatment. | Day 0 (inclusion) ; up to 4 months
  comparison of mean monthly epistaxis duration 3 months before the treatment and 3 months after the end of the treatment.

SECONDARY OUTCOMES:
Tolerance of timolol nasal spray in patients with HHT-related epistaxis | up to 7 months
  Tolerance will be evaluated by observing adverse effects and clinical examinations during the follow up period.
Efficacy on clinical criteria : epistaxis frequency . | Day 0 (inclusion) ; up to 4 months
  Comparison of number of epistaxis before and after treatment.
Efficacy on clinical criteria : biological parameters (hemoglobin and ferritin level). | Day 0 (inclusion) ; up to 4 months
  Comparison of hemoglobin and ferritin level before and after treatment.
Efficacy on clinical criteria : quality of life (SF36). | Day 0 (inclusion) ; up to 4 months
  Comparison of SF36 questionnaire before and after treatment.
Efficacy of timolol nasal spray on duration of nosebleeds for 6 months after the end of the treatment. | Day 0 (inclusion) ; up to 7 months
  Comparison of mean monthly epistaxis duration 3 months before the treatment and 6 months after the end of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Femme Mère Enfant / Service de génétique Clinique, Bron, France

REFERENCES:
- [Result] Dupuis-Girod S, Pitiot V, Bergerot C, Fargeton AE, Beaudoin M, Decullier E, Breant V, Colombet B, Philouze P, Faure F, Letievant JC. Efficacy of TIMOLOL nasal spray as a treatment for epistaxis in hereditary hemorrhagic telangiectasia. A double-blind, randomized, placebo-controlled trial. Sci Rep. 2019 Aug 19;9(1):11986. doi: 10.1038/s41598-019-48502-9. PMID 31427745
- See also: Related Info — http://www.rendu-osler.fr